CLINICAL TRIAL: NCT06269679
Title: 3D Imaging (Cone Beam Computed Tomography) Versus Orthopantomogram on the Oral Health Status at 12 Months of Patients Hospitalized for Infective Endocarditis: a Multicenter Randomized Superiority Controlled Trial.
Brief Title: CBCT vs OPT on the Oral Health Status at 12 Months of Patients Hospitalized for Infective Endocarditis.
Acronym: 3D STARS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RC23_0336
Record Dates: First submitted 2024-02-05; First posted 2024-02-21 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2024-12

CONDITIONS: Infective Endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OPT (No Intervention): Orthopantomogram = current recommended clinical examination approach (comparator procedure)
- CBCT (Experimental): Cone Beam Computed Tomography = experimental clinical examination approach (procedure under evaluation)
  Interventions: Diagnostic Test: CBCT

INTERVENTIONS:
Diagnostic Test: CBCT — Cone Beam Computed Tomography (CBCT) has a better sensitivity and sensibility to detect OIF.
  Arms: CBCT

SUMMARY:
1. Infective Endocarditis (IE) is a rare and serious disease with high morbidity and mortality; 2. Streptoccoci of oral origin are the second more frequent microorganisms responsible for IE; 3. Oral Infectious Foci (OIF) are underdetected using the current recommended clinical examination/Orthopantomogram (OPT) approach; 4. Cone Beam Computed Tomography (CBCT) has a better sensitivity and sensibility to detect OIF than OPT; 5. To date, no study has been performed to assess the potential benefit of a clinical examination/CBCT approach on the oral health status in IE patients.

Thus, conducting a randomized controlled trial is highly desirable to assess the potential impact of a clinical examination/CBCT approach on the oral health status of patients hospitalized for IE and potentially to reduce IE new episodes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients hospitalized or recently hospitalized for definite IE according to the 2015 ESC classification, naive patients for dental examination and imaging, whatever the IE responsible microorganism;
2. Patients with a stable clinical state, meaning stabilized IE patients out of the critical phase, compatible with the performance of an OPT and a CBCT;
3. Patients whose life expectancy is expected to be longer than 6 months;
4. Patients who agree to visit the dental department of the hospital to carry out OIF eradication or at his/her personal dentist;
5. Patients over 18 years old;
6. Patients affiliated to a Social Security or a health insurance scheme;
7. Patients who have given informed consent to participate to the study.

Exclusion Criteria:

1. OPT or CBCT already performed before the inclusion of the patients in the study and available for the investigator during the patient's hospitalization.
2. Medical contraindications to perform OPT or CBCT imaging;
3. Absence of microbiologic identification of the IE responsible microorganism;
4. Pregnant or breastfeeding women;
5. Patients unable to give informed consent to participate to the study (under trusteeship, guardianship and legal protection).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2028-07-18 (Estimated); Study Completion 2028-07-18 (Estimated)

PRIMARY OUTCOMES:
Superiority of CBCT | Month 12
  Number of oral infectious foci detected using orthopantomogram versus Cone Beam Computer Tomography
Superiority of CBCT | Month 12
  DFMT index comprising the number of decayed, filled and missing teeth
Superiority of CBCT | Month 12
  Number of severe periodontitis sites

SECONDARY OUTCOMES:
Diagnostic at inclusion | Day 0
  Determine the diagnostic impact of clinical examination combined with CBCT at inclusion visit (Number of OIF detected at inclusion visit through clinical examination and CBCT versus clinical examination and OPT).
Incident symptomatic OIF | Month 12
  Monitor incident symptomatic OIF occuring during the study impacting the initial personalized OIF management (Number of incident symptomatic OIF detected during the study).
Incident asymptomatic OIF | Month 12
  Monitor incident asymptomatic OIF occuring during the study i.e. OIF absent at the initial examination but identified at the ultimate visit without symptomatic episode, in patients subjected to a clinical oral examination coupled with a CBCT (Number of incident asymptomatic OIF occuring during the study i.e. OIF absent at the initial examination but detected at the ultimate visit without symptomatic episode, in patients subjected to a clinical oral examination coupled with a CBCT).
Oral hygiene | Day 0 and Month 12
  Evaluate the oral hygiene of the IE patients included in the study (Oral hygiene using the Oral Hygiene Index- Simplified score (OHI-S) at inclusion visit and at the end-of-study visit).
Follow-up habits | Day 0 and Month 12
  Evaluate the follow-up habits of the IE patients included in the study by number of dental visits per year at inclusion visit and at the end-of-study visit).
Follow-up habits | Day 0 and Month 12
  Evaluate the follow-up habits of the IE patients included in the study by number of dental brushings per day (specific questionnaire already validated in French version) at inclusion visit and at the end-of-study visit).
Oral health quality of life | Day 0 and Month 12
  Assess the oral health quality of life of the IE patients included in this study (Oral health quality of life using by the short version of the self-administrated Oral Health impact profile-14 questionnaire (OHIP-14), at inclusion visit and at the end-of-study visit).
Premature end of study | Month 12
  Analyse the patient's premature end of study (Causes of the patient's premature end of study: loss to follow-up, death, patient withdrawing consent).
Impact of dental OIF | Month 12
  Number of dental OIF detected at the end-of-study visit through clinical examination versus number of periodontal OIF detected at the inclusion visit through clinical examination.
Impact of periodontal OIF | Month 12
  Number of periodontal OIF detected at the end-of-study visit through clinical examination versus number of periodontal OIF detected at the inclusion visit through clinical examination.
Impact of mucosal OIF | Month 12
  Number of mucosal OIF detected at the end-of-study visit through clinical examination versus number of periodontal OIF detected at the inclusion visit through clinical examination.

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - CHU Bordeaux - Site Pellegrin, Bordeaux
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - HCL, Lyon
  - APHM, Marseille
  - CHRU Nancy, Nancy
  - CHU Nantes, Nantes
  - AP-HP - Site Bretonneau, Paris
  - CHU Toulouse, Toulouse
  - CHRU Tours, Tours

IPD SHARING:
Plan to Share IPD: No